CLINICAL TRIAL: NCT01460290
Title: Asenapine in the Treatment of Older Adults With Bipolar Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Martha Sajatovic, Professor of Psychiatry, University Hospitals Cleveland Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 39358
Record Dates: First submitted 2011-10-24; First posted 2011-10-26 (Estimated); Results first posted 2014-08-05 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — asenapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Asenapine (Experimental): 12-weeks of open-label asenapine treatment
  Interventions: Drug: Asenapine

INTERVENTIONS:
Drug: Asenapine — Asenapine will be administered open-label in pill form. Asenapine will be initiated at 5 mg twice a day and increased as tolerated to a maximum of 20 mg/day. It is anticipated that maximum stable dosing will be achieved by 4 weeks of treatment, although dosage may be reduced due to tolerability concerns at the discretion of the treating research psychiatrist.
  Other Names: Saphris

SUMMARY:
Objectives: The investigators propose a first-ever, prospective trial of asenapine in older adults with bipolar disorder (BD) to evaluate effects on mood symptoms, tolerability and functional/general health status. Given the dearth of treatment data on older adults with BD, findings are likely to be of substantial clinical interest, may inform larger future studies and will assist in refining bipolar treatment recommendations.

Hypotheses:

Primary: Asenapine therapy will be associated with reduced bipolar manic and depressive symptoms in older adults with BD.

Secondary: Asenapine therapy will be associated with improved functional and general health status, improved global psychopathology, and good tolerability in older adults with BD.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have type I Bipolar disorder by DSM-IV criteria confirmed on the Mini Neuropsychiatric Interview (MINI)
* Subjects must be age 60 or older
* Subjects must have sub-optimal response to current psychotropic management including at least one of the following:

  1. Behaviors and symptoms of irritability, agitation, mood lability or diminished ability to interact with others in their place of residence
  2. Diminished ability to take care of basic personal needs in their place of residence due to symptoms of BD

Exclusion Criteria:

* History of intolerance or resistance to asenapine
* Clinical diagnosis of dementia or Mini-mental state (MMSE) < 24
* History of TIA, stroke or MI within the past 12 months
* Medical illness that is the clear, underlying etiology of BD
* Unstable medical illness or condition including prolonged QT interval, which in the opinion of the study investigators, is likely to affect the outcome of the study or the subject's safety
* DSM-IV substance dependence (except nicotine or caffeine) within the past 3 months.
* Rapid cycling BD defined as 4 or more discrete mood episodes within the previous 12 months.
* At high risk for self-harm or suicide

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martha Sajatovic, M.D., Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Asenapine: 12-weeks of open-label asenapine treatment. Asenapine was administered open-label in pill form. Asenapine was initiated at 5 mg and increased as tolerated to a maximum of 20 mg/day. A control group was not used for this study.
Period: Overall Study
Arm/Group | Asenapine
Started | 15
Completed | 11
Not Completed | 4
Not completed — Adverse Event | 3
Not completed — Elevated liver function | 1

BASELINE CHARACTERISTICS:
Groups:
- Asenapine: 12-weeks of open-label asenapine treatment
  Asenapine was administered open-label in pill form. Asenapine was initiated at 5 mg/day and increased as tolerated to a maximum of 20 mg/day. A control group was not used for this study.
Arm/Group | Asenapine
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.6 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Depressive Symptoms as Measured by the Hamilton Depression Rating Scale (HAM-D)
Description: The minimum possible score is 0 and the maximum score is 52. A higher score implies a worse condition.
Time Frame: Baseline and 12 weeks
Population: Participants with baseline HAM-D score of 8 or greater were analyzed. Last Observational Carried Forward (LOCF).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Asenapine
Number analyzed (Participants) | 11
units on a scale
  Baseline HAM-D | 17.5 (4.8)
  12 Week HAM-D | 10.3 (6.3)

2. Primary Outcome: Change in Manic Symptoms as Measured by the Young Mania Rating Scale (YMRS)
Description: The minimum possible score is 0 and the maximum score is 60. A higher score implies a worse condition.
Time Frame: Baseline and 12 weeks
Population: Participants with a baseline YMRS score of 12 or greater were analyzed. LOCF
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Asenapine
Number analyzed (Participants) | 5
units on a scale
  Baseline YMRS | 27.9 (4.4)
  12 Week YMRS | 18.1 (14.2)

3. Secondary Outcome: Change in Global Psychopathology as Measured by the Clinical Global Impression Scale for Use in Bipolar Illness (CGI-BP)
Description: The minimum possible score is 1 and the maximum score is 7. A higher score implies a worse condition.
  The CGI-BP has three scores - Mania Severity, Depression Severity, and Overall Bipolar Illness Severity.
Time Frame: Baseline and 12 weeks
Population: Intention To Treat (ITT) and LOCF
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Asenapine
Number analyzed (Participants) | 15
units on a scale
  Baseline Overall Severity | 4.4 (1.0)
  12 Week Overall Severity | 2.2 (1.0)
  Baseline Mania Severity | 2.7 (1.7)
  12 Week Mania Severity | 1.9 (1.1)
  Baseline Depression Severity | 3.6 (1.5)
  12 Week Depression Severity | 1.7 (0.7)

4. Secondary Outcome: Change in Perception of Physical Health as Measured by the Short Form General Health Survey (SF-12)
Description: The minimum possible score is 1 and the maximum score is 99. A higher score implies a better perceived condition.
Time Frame: Baseline and 12 weeks
Population: ITT and LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Asenapine
Number analyzed (Participants) | 15
units on a scale
  Baseline on Physical Health Subscale of SF-12 | 46.8 (11.3)
  12 week on Physical Health Subscale of SF-12 | 46.4 (12.1)

5. Secondary Outcome: Change in Perception of Mental Health as Measured by the Short Form General Health Survey (SF-12)
Description: The minimum possible score is 1 and the maximum score is 99. A higher score implies a better perceived condition.
Time Frame: Baseline and 12 weeks
Population: ITT and LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Asenapine
Number analyzed (Participants) | 15
units on a scale
  Baseline Mental Health Subscore of SF-12 | 38.7 (15.3)
  12 Week Mental Health Subscore of SF-12 | 43.1 (13.1)

6. Secondary Outcome: Change in Depressive Symptoms as Measured by the Montgomery Asberg Depression Rating Scale (MADRS)
Description: The minimum possible score is 0 and the maximum score is 60. A higher score implies a worse condition.
Time Frame: Baseline and 12 weeks
Population: Participants with a baseline MADRS score of 16 or greater were analyzed. LOCF
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Asenapine
Number analyzed (Participants) | 9
units on a scale
  Baseline MADRS | 27.9 (4.4)
  12 Week MADRS | 18.1 (14.2)

7. Secondary Outcome: Change in Bipolar Disorder Symptoms as Measured by the Brief Psychiatric Rating Scale (BPRS)
Description: The minimum possible score is 18 and the maximum score is 126. A higher score implies a worse condition.
Time Frame: Baseline and 12 weeks
Population: ITT and LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Asenapine
Number analyzed (Participants) | 15
units on a scale
  Baseline BPRS | 35.1 (9.2)
  12 Week BPRS | 28.6 (9.4)

8. Secondary Outcome: Change in Cognitive Status as Measured by the Stroop Task
Description: The Stroop evaluates patients for cognitive functioning. Patients are to read words aloud or name colors as quickly as possible in a 45-second period. The measure contains three tasks, each associated with a subscale as follows: Word, Color, and Color-Word. Each subscale contains 100 items. The raw score range for each of the subscales is 0-100. Each raw subscale score is converted to a T-Score. The possible T-Score range for the Word subscale is 15 to 85. The possible T-Score range for the Color subscale is 8 to 92. The possible T-Score range for the Color-Word subscale is 3 to 98. Higher scores on the subscales indicate better cognitive functioning. Subscales are scored independently and are not added to produce a total score.
Time Frame: Baseline and 12 weeks
Population: Participants who completed cognitive scales at baseline and at Week 12 visit were analyzed.
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Asenapine
Number analyzed (Participants) | 9
T-Score
  Baseline Word Subscale | 75.7 (12.0)
  12 Week Word Subscale | 75.9 (11.5)
  Baseline Color Subscale | 53.6 (9.2)
  12 Week Color Subscale | 58.6 (7.7)
  Baseline Color-Word Subscale | 30.3 (11.4)
  12 Week Color-Word Subscale | 30.6 (10.1)

9. Secondary Outcome: Change in Cognitive Status as Measured by the Trail Making Test
Description: The Trails test is a measure of cognitive functioning. The measure consists of two parts: A and B. In part A, participants are asked to draw a trail connecting a series of numbers in sequential order. In Part B, participants are asked to draw a trail connecting a combination of letters and numbers. The time taken to complete each task is noted as the score (e.g., 78 seconds). For Trails A, there is no upper limit on the score, as subjects are given as much time as is needed for them to complete the task. Higher scores indicate poorer cognitive functioning. In Trails B, the task is timed with an upper limit of five minutes. If, at four minutes, it is determined that the subject will not likely complete the task in the time allotted, then the task can be called off. Higher scores indicate poorer cognitive functioning.
Time Frame: Baseline and 12 weeks
Population: Participants who completed cognitive scales at baseline and at Week 12 visit were analyzed.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Asenapine
Number analyzed (Participants) | 9
seconds
  Baseline Trails - Part A | 57.7 (30.9)
  12 Week Trails - Part A | 47.3 (10.4)
  Baseline Trails - Part B | 189.0 (103.8)
  12 Week Trails - Part B | 126.3 (52.4)

10. Secondary Outcome: Change in Cognitive Status as Measured by the Hopkins Verbal Learning Test (HVLT)
Description: Evaluates cognitive functioning across domains: recall, delayed recall, retention, recognition (each scored separately). The scores given are titled: recall score, delayed recall score, retention score, recognition discrimination index. Total Recall score = items correctly recalled (0-36). Delayed Recall score = items correctly recalled following delay (0-12). Retention score = percent items recalled that were also recalled after delay (0-100). The Recognition Discrimination score = true positives minus false positives (0-12). Recall task has 12 words and involves to recall of words after all of them are read aloud to the patient. Delayed recall tasks involves the same twelve words, except recall is tasked after a 20-25 minute delay. Recognition task has 24 words. Patient evaluated on how many from original list he or she is able to recognize. Higher scores = better outcomes.
  Total recall scores appear in this entry below.
Time Frame: Baseline and 12 weeks
Population: Participants who completed cognitive scales at baseline and at Week 12 visit were analyzed.
Measure: Mean (Standard Deviation); unit: correctly recalled items
Arm/Group | Asenapine
Number analyzed (Participants) | 9
correctly recalled items
  Baseline HVLT Total Recall | 15.8 (5.7)
  12 Week HVLT Total Recall | 18.2 (5.4)

11. Secondary Outcome: Change in Cognitive Status as Measured by the Dementia Rating Scale (DRS)
Description: The DRS contains items that evaluate cognitive function across 5 subscales: attention, initiation/perseveration, construction, conceptualization, and memory. Subscale raw score ranges are: attention (0-37), initiation/perseveration (0-37), construction (0-6), conceptualization (0-39), and memory (0-25). Raw subscale scores are added for a total raw score with range 0-144. For each raw subscale score, scaled scores are looked up from a battery of 13 tables. Age of the participant determines which table is to be used. Total raw subscale score also has its own scaled score in the tables. In addition to use in determining scaled scores for each of the subscales, these tables are used to look up the scaled score for the total raw score. The tables are contained in the article Robust and Expanded Norms for the Dementia Rating Scale (Pedraza, Lucas, et al. 2010); Archives of Clinical Neuropsychology 25; 347-358. Higher scores, raw and scaled, indicate better cognitive functioning.
Time Frame: Baseline and 12 weeks
Population: Participants who completed cognitive scales at baseline and at Week 12 visit were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Asenapine
Number analyzed (Participants) | 9
units on a scale
  Baseline DRS | 131.2 (6.6)
  12 Week DRS | 135.6 (6.6)

12. Secondary Outcome: World Health Organization Disability Assessment Scale (WHO-DAS)
Description: The WHO-DAS II is used to assess patients for difficulties that they experience due to health conditions. Six subscales are represented which cover the following domains: Getting Around (range 1-10), Self Care (range 1-10), Life Activities (range 1-20), Understand/Communicate (range 1-10), Participation in Society (range 1-10), and Getting Along with People (range 1-10). Lower scores represent more positive outcomes, while higher scores represent worse outcomes. Total summary scores were not computed for our analyses and is optional for the measure.
Time Frame: 12 weeks
Population: ITT and LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Asenapine
Number analyzed (Participants) | 15
units on a scale
  Baseline WHO-DAS Getting Around Subscale | 4.3 (2.7)
  12 Week WHO-DAS Getting Around Subscale | 4.7 (2.9)
  Baseline WHO-DAS Self Care Subscale | 2.6 (1.3)
  12 Week WHO-DAS Self Care Subscale | 2.4 (0.7)
  Baseline WHO-DAS Life Activities Subscale | 9.1 (4.9)
  12 Week WHO-DAS Life Activities Subscale | 7.1 (3.5)
  Baseline WHO-DAS Understand/Communicate Subscale | 3.6 (1.8)
  12 Week WHO-DAS Understand/Communicate Subscale | 3.1 (1.2)
  Baseline WHO-DAS Participation in Society Subscale | 4.3 (2.6)
  12 Week WHO-DAS Participation in Society Subscale | 3.8 (2.0)
  Baseline WHO-DAS Getting Along w/ People Subscale | 3.0 (1.5)
  12 Week WHO-DAS Getting Along w/ People Subscale | 2.9 (1.9)

13. Secondary Outcome: Barnes Drug-induced Akathisia Rating Scale (BARS)
Description: This scale is used to measure the presence of akathisia, as may result from use of certain psychotropic medications. The scale contains four items and the score for each item is added to produce the total score. Total scores range from 0 to 14. Higher scores indicate more adverse outcomes.
Time Frame: Baseline and 12 weeks
Population: ITT and LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Asenapine
Number analyzed (Participants) | 15
units on a scale
  Baseline BARS | 0.0 (0.0)
  12 Week BARS | 0.1 (0.5)

14. Secondary Outcome: Assessment of Motor Control Abnormality as Measured by the Simpson Angus Scale (SAS)
Description: The Simpson-Angus Scale is used to monitor for neurological and musculoskeletal side effects that may be a result of certain psychotropic medications. The scale consists of 10 questions which each can be rated on a scale of 0 to 4. Scores for each item are added to produce a total score. The highest possible total score is 40. Higher scores indicate more adverse outcomes.
Time Frame: Baseline and 12 weeks
Population: ITT and LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Asenapine
Number analyzed (Participants) | 15
units on a scale
  Baseline SAS | 0.4 (0.8)
  12 Week SAS | 0.5 (0.7)

15. Secondary Outcome: Change in Cognitive Status as Measured by the Hopkins Verbal Learning Test (HVLT)
Description: Evaluates cognitive functioning across domains: recall, delayed recall, retention, recognition (each scored separately). The scores given are titled: recall score, delayed recall score, retention score, recognition discrimination index. Total Recall score = items correctly recalled (0-12). Delayed Recall score = items correctly recalled following delay (0-12). Retention score = percent items recalled that were also recalled after delay (0-100). The Recognition Discrimination score = true positives minus false positives (0-12). Recall task has 12 words and involves to recall of words after all of them are read aloud to the patient. Delayed recall tasks involves the same twelve words, except recall is tasked after a 20-25 minute delay. Recognition task has 24 words. Patient evaluated on how many from original list he or she is able to recognize. Higher scores = better outcomes.
  Delayed recall scores appear in this entry below.
Time Frame: Baseline and 12 weeks
Population: Participants who completed cognitive scales at baseline and at Week 12 visit were analyzed.
Measure: Mean (Standard Deviation); unit: correctly recalled items
Arm/Group | Asenapine
Number analyzed (Participants) | 9
correctly recalled items
  Baseline HVLT Delayed Recall | 5.2 (3.0)
  12 Week HVLT Delayed Recall | 5.3 (2.7)

16. Secondary Outcome: Change in Cognitive Status as Measured by the Hopkins Verbal Learning Test (HVLT)
Description: Evaluates cognitive functioning across domains: recall, delayed recall, retention, recognition (each scored separately). The scores given are titled: recall score, delayed recall score, retention score, recognition discrimination index. Total Recall score = items correctly recalled (0-12). Delayed Recall score = items correctly recalled following delay (0-12). Retention score = percent items recalled that were also recalled after delay (0-100). The Recognition Discrimination score = true positives minus false positives (0-12). Recall task has 12 words and involves to recall of words after all of them are read aloud to the patient. Delayed recall tasks involves the same twelve words, except recall is tasked after a 20-25 minute delay. Recognition task has 24 words. Patient evaluated on how many from original list he or she is able to recognize. Higher scores = better outcomes.
  Retention scores appear in this entry below.
Time Frame: Baseline and 12 weeks
Population: Participants who completed cognitive scales at baseline and at Week 12 visit were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of items
Arm/Group | Asenapine
Number analyzed (Participants) | 9
percentage of items
  Baseline HVLT Retention | 73.9 (32.7)
  12 Week HVLT Retention | 71.8 (34.4)

17. Secondary Outcome: Change in Cognitive Status as Measured by the Hopkins Verbal Learning Test (HVLT)
Description: Evaluates cognitive functioning across domains: recall, delayed recall, retention, recognition (each scored separately). The scores given are titled: recall score, delayed recall score, retention score, recognition discrimination index. Total Recall score = items correctly recalled (0-12). Delayed Recall score = items correctly recalled following delay (0-12). Retention score = percent items recalled that were also recalled after delay (0-100). The Recognition Discrimination score = true positives minus false positives (0-12). Recall task has 12 words and involves to recall of words after all of them are read aloud to the patient. Delayed recall tasks involves the same twelve words, except recall is tasked after a 20-25 minute delay. Recognition task has 24 words. Patient evaluated on how many from original list he or she is able to recognize. Higher scores = better outcomes.
  Recognition Discrimination Index appears in this entry below
Time Frame: Baseline and 12 weeks
Population: Participants who completed cognitive scales at baseline and at Week 12 visit were analyzed.
Measure: Mean (Standard Deviation); unit: number of items
Arm/Group | Asenapine
Number analyzed (Participants) | 9
number of items
  Baseline HVLT Recognition Discrimation Index | 8.6 (2.5)
  12 Week HVLT Recognition Discrimination Index | 9.6 (2.0)

ADVERSE EVENTS:
Arm/Group | Asenapine
Serious Adverse Events (participants affected / at risk) | 3/15
Other Adverse Events (participants affected / at risk) | 13/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asenapine (N=15)
emergence of manic symptoms (Psychiatric disorders) | 1 (1) — Determined to be possibly study related
recurrence of suicidal ideation (Psychiatric disorders) | 1 (1) — Occurred in the context of tooth abscess Determined to be not study related
reported dizziness/refusal to take additional mood stabilizer (Psychiatric disorders) | 1 (1) — occurred after taking a single dose of asenapine in an individual with euphoric mania Determined to be not study related
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asenapine (N=15)
elevated liver functions (Hepatobiliary disorders) | 1 (1) — Resolved with drug discontinuation. Determined to be possibly related to study drug
gastrointestinal discomfort (Gastrointestinal disorders) | 5 (5)
restlessness (General disorders) | 2 (2)
tremors (General disorders) | 2 (2)
cognitive difficulties (General disorders) | 2 (2)
sluggishness/sedation (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No